CLINICAL TRIAL: NCT01470365
Title: Phase I Study of Pulsed Low Dose Rate Reirradiation Delivered With 3DCRT/IMRT for Palliation of Recurrent Tumors
Brief Title: 3-Dimensional Conformal Radiation Therapy or Intensity-Modulated Radiation Therapy in Treating Patients With Recurrent Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OER-RT-042; NCI-2011-03311 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB#11-044/OER-RT-042 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2011-11-03; First posted 2011-11-11 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation therapy) (Experimental): Patients undergo 3-dimensional CRT or IMRT QD, 5 days a week for 10-30 days. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: quality-of-life assessment; Radiation: intensity-modulated radiation therapy; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Radiation: 3-dimensional conformal radiation therapy — Undergo 3-dimensional CRT
  Other Names: 3D conformal radiation therapy; 3D-CRT

SUMMARY:
This phase I trial studies the side effects and best dose of 3-dimensional conformal radiation therapy (CRT) or intensity-modulated radiation therapy (IMRT) in treating patients with recurrent tumors. Radiation therapy (RT) uses high energy x rays to kill tumor cells. Palliative radiation therapy may help patients with recurrent tumors live more comfortably.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of reirradiation with the pulsed low dose rate technique.

SECONDARY OBJECTIVES:

I. To investigate the dosimetric tolerance of normal structures to reirradiation with the pulsed low dose rate technique.

II. To determine the palliative efficacy and quality of life in patients treated on this protocol.

III. To determine duration of response and time to progression.

OUTLINE: This is a dose-escalation study.

Patients undergo 3-dimensional CRT or IMRT once daily (QD), 5 days a week for 10-30 days. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every month for 6 months and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed malignancy
* Patients must have recurrent or metastatic tumor located within a previously irradiated field
* Tumor within the irradiated field is negatively impacting patient's quality of life or threatening catastrophic complication if left untreated as determined by the treating physician
* Patient is not a candidate for, or has not demonstrated a significant local response to chemotherapy, biologic, hormonal ,or other therapies
* Patient is not a surgical candidate or tumor is not surgically resectable, as documented by surgical oncologist
* Information on previous radiation treatment, including total dose and fractionation must be available; additional information including radiation fields and dose-volume-histogram or isodose lines is preferable
* Tumor sites eligible for inclusion on this protocol include thorax, abdomen, and pelvis
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in the previously irradiated field
* Women of childbearing potential must be non-pregnant (negative pregnancy test within 72 hours prior to radiation simulation, postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential) and nonlactating, and men and women must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 3 months after therapy completed
* Eastern Cooperative Oncology Group (ECOG) performance status determined to be between 0 and 3
* Absolute neutrophil count (ANC) >= 1,500/ul
* Platelets (PLT) >= 75,000/ul
* Subjects must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy to the reirradiation target within 4 weeks prior to entering the study
* Concurrent chemotherapy or biologic therapy
* A history of ataxia telangiectasia or other documented history of radiation hypersensitivity
* Scleroderma or active connective tissue disease
* For abdominal or pelvic irradiation: active inflammatory bowel disease
* Serious, active infections requiring treatment with intravenous (IV) antibiotics
* Uncontrolled intercurrent illness including, but not limited to, or psychiatric illness/social situations that would limit compliance with study requirements
* Reirradiation targets located within the head, neck, or brain are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11-03 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
MTD of reirradiation with the pulsed low dose rate technique | Up to 30 days
  Defined as the dose level closest to, but not over that which is predicted to result in a dose limiting toxicity (DLT) rate of 20%, the target toxicity rate. Graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. A DLT is a grade >= 4 acute or grade >= 3 late toxicity of an organ system within the reirradiation field in the following categories: skin or subcutaneous tissues, gastrointestinal, hepatobiliary, nervous system, renal and urinary, reproductive system, vascular, or respiratory, thoracic and mediastinal disorders.

SECONDARY OUTCOMES:
Palliative efficacy in terms of quality of life and pain levels | Up to 3 years
  Assessed using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 15 Palliative (QLQ-C15-PAL) and the Numeric Pain Scale. The mean and standard deviation will be estimated at each time point.
Duration of response | Up to 3 years
  Measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Assessed using the RECIST 1.1 criteria. Estimated using Kaplan-Meier curves.
Time to progression | Up to 3 years
  Assessed using the RECIST 1.1 criteria. Estimated using Kaplan-Meier curves.

CONTACTS AND LOCATIONS:
Overall Officials: C-M Charlie Ma, PhD, Principal Investigator — Fox Chase Cancer Center; Josphua Meyer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States